CLINICAL TRIAL: NCT06560268
Title: Effects of Different Fresh Gas Flows on Emergence Agitation and Anesthetic Agent Consumption in Children Undergoing Strabismus Surgery
Brief Title: Low Flow Anesthesia in Children Undergoing Strabismus Surgery
Acronym: LFA in child
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Feride Karacaer, Associate Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3/21.03.2024
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Low Flow Anesthesia; Sevoflurane; Strabismus; Emergence Delirium
Keywords: emergence agitation; strabismus; children; low flow anesthesia
MeSH Terms: conditions — Strabismus; Emergence Delirium | interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High flow anesthesia (Experimental): Group I; After the laryngeal mask is placed, ventilation will be performed with FGF= 4 l/min, Sevoflurane vaporizer setting will be 2.5-3%. When the patients reach 1 MAC Sevoflurane, FGF will be reduced to 2 l/min.
  In Group I, the Sevoflurane vaporizer will be turned off at the end of the operation and FGF will be increased to 10 l/min.
  Interventions: Drug: Sevoflurane; In our study, the effects of sevoflurane in different FGFs administered in children undergoing strabismus surgery on EA and anesthetic agent consumption will be investigated.
- Low flow anesthesia (Experimental): Group II; After the laryngeal mask is placed, ventilation will be performed with FGF= 4 l/min, Sevoflurane vaporizer setting will be 2.5-3% and when the patients reach 1 MAC, FGF= 0.5 l/min will be reduced.
  In Group II, the Sevoflurane vaporizer will be turned off 10 minutes before the end of the operation and FGF will continue as 0.5 l/min until the end of the operation.
  Interventions: Drug: Sevoflurane; In our study, the effects of sevoflurane in different FGFs administered in children undergoing strabismus surgery on EA and anesthetic agent consumption will be investigated.
- Low flow wash-in period (Experimental): Group III; After the laryngeal mask is placed, ventilation will be performed with FGF= 1 l/min, Sevoflurane vaporizer setting will be 8%, inhaled sevoflurane concentration (Fisevo) will be gradually reduced to < 4%. When the children reach 1 MAC sevoflurane, TGA= 0.5 l/min will be reduced.
  In Group III, the sevoflurane vaporizer will be turned off 10 minutes before the end of the operation and FGF will continue as 0.5 l/min until the end of the operation.
  Interventions: Drug: Sevoflurane; In our study, the effects of sevoflurane in different FGFs administered in children undergoing strabismus surgery on EA and anesthetic agent consumption will be investigated.

INTERVENTIONS:
Drug: Sevoflurane; In our study, the effects of sevoflurane in different FGFs administered in children undergoing strabismus surgery on EA and anesthetic agent consumption will be investigated. — Low-flow anaesthesia is generally adminstered as nitrogen wash-out, a period of higher flow rate in combination with a high vaporizer setting for initial saturation, and subsequent reduction of fresh gas flow and adjustment of the vaporizer to maintain the desired end-tidal anesthetic agent concentration (Etaa).In the initial wash-in phase, the vaporizer setting is adjusted to 6% for desflurane and 2.5-3% for sevoflurane, with FGF=4 L/min, until the Etaa concentration is 1-1.3 MAC. In another method, the vaporizer setting is adjusted to 12-18% for desflurane and 6-8% for sevoflurane, with FGA=1 L/min. Reducing the FGF during the wash-in period prevents unnecessary depth of anesthesia and reduces the consumption of inhalational anesthetics. In LFA using minimal FGF (250-500 mL/min), if the vaporizer is turned off 10-15 min before the end of the operation and the FGF is not changed, the inhaled anesthetic agent concentration gradually and slowly decreases to zero.

SUMMARY:
Emergence agitation (EA) involves restlessness, disorientation, excitation, non-purposeful movement, inconsolability, thrashing, and incoherence during early recovery from general anesthesia. Sevoflurane and desflurane have increased the incidence of EA in children. A proposed explanation for this is that sevoflurane and desflurane cause differential recovery rates in brain function, due to differences in clearance of inhalational anesthetics from the central nervous system; whereas audition and locomotion recover first, cognitive function recovers later, resulting in EA. Low-flow anaesthesia (LFA) occurs when the fresh gas flow (FGF) is significantly lower than the patient's minute volume. In a low-flow system, the recirculated fraction should amount to at least 50% after carbon dioxide (CO2) absorption.In LFA using minimal FGF (250-500 mL/min), if the vaporizer is turned off 10-15 minutes before the end of the operation and the FGF is not changed, the inhaled anesthetic agent concentration gradually and slowly decreases to zero and the inhaled agent consumption decreases even more. In a study conducted on infants undergoing cleft lip-palate surgery, it was shown that the incidence of postoperative agitation were statistically lower in infants who administered 0.5 L/min FGF.

Strabismus surgery is one of the most frequently performed ophthalmologic operations in children and is associated with moderate postoperative pain and a high incidence of EA (40-86%). The incidence of EA after strabismus surgery is high, especially due to visual disturbances; however, the pathogenesis of this condition remains unclear. In our study, the effects of different FGFs administered in children undergoing strabismus surgery on EA and anesthetic agent consumption will be investigated.

DETAILED DESCRIPTION:
Emergence agitation (EA) involves restlessness, disorientation, excitation, non-purposeful movement, inconsolability, thrashing, and incoherence during early recovery from general anesthesia. The incidence of EA varies, from approximately 0.25% to 90.5%, with age, assessment tool used, definitions, anesthetic techniques, type of surgery, and time of EA assessment during recovery. The clinical consequences of EA are similarly varied. It is typically short lived and resolves spontaneously, and its clinical consequences are often considered minimal. However, it may have clinically significant consequences, such as injury to the affected patient or their medical staff, falling out of bed, bleeding at the surgical site, accidental removal of drains or intravenous catheters, unintended extubation, respiratory depression, and increasing medical care costs.

Sevoflurane and desflurane have increased the incidence of EA in children. A proposed explanation for this is that sevoflurane and desflurane cause differential recovery rates in brain function, due to differences in clearance of inhalational anesthetics from the central nervous system; whereas audition and locomotion recover first, cognitive function recovers later, resulting in EA. In addition, studies on pediatric patients have found that being awakened rapidly by unfamiliar healthcare personnel in an unfamiliar operating room environment is a potential risk factor for EA. Rapid clearance of anesthetic agents from subcortical structures (locus coeruleus and amygdala) before the cerebral cortex and rapid recovery have been suggested as a causal factor for EA. Therefore, methods to reduce the incidence of EA aim to reduce the concentration difference between cortical and subcortical areas by slowing down the elimination of inhaled anesthetic agents.

Low-flow anaesthesia (LFA) occurs when the fresh gas flow (FGF) is significantly lower than the patient's minute volume. In a low-flow system, the recirculated fraction should amount to at least 50% after carbon dioxide (CO2) absorption. There are various techniques for the introduction of the inhaled anesthetic. In general, they all follow the same sequence: nitrogen wash-out, a period of higher flow rate in combination with a high vaporizer setting for initial saturation, and subsequent reduction of fresh gas flow and adjustment of the vaporizer to maintain the desired end-tidal anesthetic agent concentration (Etaa). The wash-in period (saturation of the central nervous system area where the inhaled agent is effective) depends on the initial FGF and the vaporizer setting. In the initial wash-in phase, the vaporizer setting is adjusted to 6% for desflurane and 2.5-3% for sevoflurane, with FGF = 4 L/min, until the Etaa concentration is 1-1.3 MAC. In another method, the vaporizer setting is adjusted to 12-18% for desflurane and 6-8% for sevoflurane, with FGF = 1 L/min. Reducing the FGF during the wash-in period prevents unnecessary depth of anesthesia and reduces the consumption of inhalational anesthetics. The wash-in, i.e., the saturation of the gaseous compartment, is dependent on the initial fresh gas flow and the vaporizer setting. Reducing FGF from 4 to 1 L/min reduces inhalation anesthetic consumption by 45.3% (desflurane) and 51.8% (sevoflurane), respectively. In parallel, there is a significant reduction in CO2e emissions and anesthesia costs per minute of approximately 45-50%. When the Etaa concentration is 1-1.3 MAC, the maintenance period is started with a FGF between 0.25-1 L/min. In LFA using minimal FGF (250-500 mL/min), if the vaporizer is turned off 10-15 minutes before the end of the operation and the FGF is not changed, the inhaled anesthetic agent concentration gradually and slowly decreases to zero and the inhaled agent consumption decreases even more (4-5). In a study conducted on infants undergoing cleft lip-palate surgery, it was shown that the incidence of postoperative agitation were statistically lower in infants who administered 0.5 L/min FGF.

Strabismus surgery is one of the most frequently performed ophthalmologic operations in children and is associated with moderate postoperative pain and a high incidence of EA (40-86%). The incidence of EA after strabismus surgery is high, especially due to visual disturbances; however, the pathogenesis of this condition remains unclear. In our study, the effects of different FGFs administered in children undergoing strabismus surgery on EA and anesthetic agent consumption will be investigated.

METHOD 150 patients aged 3-10 years undergoing strabismus surgery will be included in the study. Patients will be randomly divided into three groups. Using a 4-point scale, preoperative agitation will be evaluated in the reception area and then, 0.05 mg/kg intravenous (iv) midazolam will be administered for premedication.

For anesthesia induction, all patients will be administered 3 mg/kg propofol and 0.5 mg/kg rocuronium and mechanical ventilation will be performed with a laryngeal mask. A tidal volume of 6-8 ml/kg will be applied and end-tidal CO2 will be maintained between 30-35 mmHg. After induction, all children will be administered 1 μg/kg fentanyl IV. In all patients, the sevoflurane concentration (in the O2 and air mixture) will be titrated between MAC= 1-1.3 throughout the operation, keeping BIS= 40-60 and baseline hemodynamic changes between ±20%. The inspiratory oxygen concentration (FiO2) alarm lower limit will be set to 30% in all patients.

Patients will be randomly divided into 3 groups:

Group I; After the laryngeal mask is placed, ventilation will be performed with FGF= 4 l/min, vaporizer setting will be 2.5-3%. When the patients reach 1 MAC, FGF will be reduced to 2 l/min.

Group II; After the laryngeal mask is placed, ventilation will be performed with FGF= 4 l/min, vaporizer setting will be 2.5-3% and when the patients reach 1 MAC, FGF= 0.5 l/min will be reduced.

Group III; After the laryngeal mask is placed, ventilation will be performed with FGF= 1 l/min, vaporizer setting will be 8%, inhaled sevoflurane concentration (Fisevo) will be gradually reduced to <4%. When the children reach 1 MAC, FGF= 0.5 l/min will be reduced.

In Group I, the vaporizer will be turned off at the end of the operation and FGF will be increased to 10 l/min.

In Group II and III, the vaporizer will be turned off 10 minutes before the end of the operation and FGF will continue as 0.5 l/min until the end of the operation.

All patients will be assessed by an anesthesiologist, who is unaware of the study protocol, at postoperative 5, 10, 15, 30 and 45. minutes and at 2 hours using the 5-point Emergence Agitation Scale and the Pediatric Anesthesia Emergence Delirium (PAED) in the postoperative recovery unit. Postoperative pain will be assessed using the Children's Hospital of Eastern Ontario Pain Scale (CHEOPS). If the patient's PAED score is ≥16, iv fentanyl (1 μg/kg) will be administered. Postoperative adverse events including laryngospasm, desaturation (SpO2<95%), nausea and vomiting will also be recorded. In the recovery unit, children with a modified Aldrete anesthesia discharge score >9 will be transferred to the ward.

ELIGIBILITY:
Inclusion Criteria:

* 3-10 years old children with strabismus

Exclusion Criteria:

* Mental retardation
* Cardiovascular disease
* Serebrovasculay disease
* Renal disease
* Hepatic disease
* Pulmonary disease

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2024-11-04 (Estimated); Primary Completion 2025-06-04 (Estimated); Study Completion 2025-07-04 (Estimated)

PRIMARY OUTCOMES:
Emergence agitation | At postoperative 5th, 10th, 15th, 30th, 45th min and 2 hour
  Comparison of emergence agitation rates between groups.

SECONDARY OUTCOMES:
Sevoflurane consumption | İntraoperative period
  Effects of different fresh gas flows on sevoflurane consumption

CONTACTS AND LOCATIONS:
Overall Officials: Feride Karacaer, Assoc Prof, Study Director — Cukurova University

REFERENCES:
- [Background] Sripriya R, Ravindran C, Murugesan R. Comparison of recovery characteristics with two different washout techniques of desflurane anaesthesia: A randomised controlled trial. Indian J Anaesth. 2020 Sep;64(9):756-761. doi: 10.4103/ija.IJA_623_20. Epub 2020 Sep 1. PMID 33162569
- [Background] Brattwall M, Warren-Stomberg M, Hesselvik F, Jakobsson J. Brief review: theory and practice of minimal fresh gas flow anesthesia. Can J Anaesth. 2012 Aug;59(8):785-97. doi: 10.1007/s12630-012-9736-2. Epub 2012 Jun 1. PMID 22653840
- [Background] Rubsam ML, Kruse P, Dietzler Y, Kropf M, Bette B, Zarbock A, Kim SC, Honemann C. A call for immediate climate action in anesthesiology: routine use of minimal or metabolic fresh gas flow reduces our ecological footprint. Can J Anaesth. 2023 Mar;70(3):301-312. doi: 10.1007/s12630-022-02393-z. Epub 2023 Feb 22. PMID 36814057
- [Background] Yang Y, Song T, Wang H, Gu K, Ma P, Ma X, Zhao J, Li Y, Zhao J, Yang G, Yan R. Comparison of two different sevoflurane expelling methods on emergence agitation in infants following sevoflurane anesthesia. Int J Clin Exp Med. 2015 Apr 15;8(4):6200-5. eCollection 2015. PMID 26131225
- [Background] Aouad MT, Nasr VG. Emergence agitation in children: an update. Curr Opin Anaesthesiol. 2005 Dec;18(6):614-9. doi: 10.1097/01.aco.0000188420.84763.35. PMID 16534301
- [Result] Voepel-Lewis T, Malviya S, Tait AR. A prospective cohort study of emergence agitation in the pediatric postanesthesia care unit. Anesth Analg. 2003 Jun;96(6):1625-1630. doi: 10.1213/01.ANE.0000062522.21048.61. PMID 12760985